CLINICAL TRIAL: NCT04223674
Title: Serological Screen and Treat Trial for P. Vivax: a Proof-of-concept Trial in Western Indonesia
Brief Title: Serological Screen and Treat Trial for Plasmodium Vivax
Acronym: SSAT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Indonesia University (Other)
Collaborators: Eijkman Institute for Molecular Biology (Other); Oxford University Clinical Research Unit Indonesia (Other); Walter and Eliza Hall Institute of Medical Research (Other); Rumah Sakit Umum Daerah Mimika (Unknown); Universitas Sumatera Utara (Other)
Responsible Party: Principal Investigator, Inge Sutanto, Professor, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 19-09-1129
Record Dates: First submitted 2020-01-03; First posted 2020-01-10 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Malaria, Vivax
Keywords: serology; screen; treat; recurrent; vivax
MeSH Terms: conditions — Malaria, Vivax; Recurrence

STUDY DESIGN:
Intervention Model Description: This study evaluates an experimental serological diagnostic technique intended to identify people at high risk of having dormant malaria parasites in their liver.
  960 children living in western Indonesia will be individually randomised to the experimental serologic test or routine care.
  Children in the serological diagnosis arm will be screened for the presence of antibodies to a previously validated panel of malaria antigens optimized for sensitivity to infection during the prior 9 months. Furthermore, they also will be screened by microscopy. If positive by either test, they will be treated for that malaria infection.
  Children assigned to routine care will be screened by microscopic examination and treated when they show or have history of symptoms in the last 3 days.
  After initial screening and treating according to diagnostic technique, all children will be actively followed for 9 months with PCR detection every 4 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Serological screen and treat (Experimental): Children who screened with sero test and microscopy. A 7-day high dose PQ will be provided for those with Pv seropositive regardless of their symptoms and symptomatic children with microscopic Pv/Po positive.
  Interventions: Diagnostic Test: Serological screen and treat
- Routine care (No Intervention): Children who screened with sero test and microscopy. A 7-day high dose PQ will be provided only for symptomatic children with microscopic Pv/Po positive.

INTERVENTIONS:
Diagnostic Test: Serological screen and treat — Multi-antigen sero-diagnostic test for measurement of P. vivax antibodies in plasma from finger stick as a means to detect hypnozoite carriers for treatment
  Arms: Serological screen and treat

SUMMARY:
This is a clinical trial to evaluate an experimental serological diagnostic technique intended to identify people at high risk of having dormant malaria parasites in their liver. The study is designed to evaluate the efficacy of serological screening vs. routine care for the prevention of recurrent P. vivax infections. A total of 960 schoolchildren will be randomized into the interventional or control arm.

DETAILED DESCRIPTION:
This is a randomized controlled trial to evaluate an experimental serological diagnostic technique intended to identify people at high risk of having dormant malaria parasites in their liver. The study is designed to show a superiority of SSAT vs. routine care for the prevention of recurrent P. vivax infections. With the estimated prevalence of 20%, the investigators will have a power of >90% to detect a significant difference with the sample size of 350 children per group. The investigators will recruit 480 children per group to anticipate subject loss due to exclusion and drop out.

After obtaining informed consent from their parents/legal guardians, 800 schoolchildren living in Batubara regency, North Sumatra, Indonesia, will be individually randomized to intervention (SSAT) or control (routine care) group. During enrollment, all participants will be tested with Pv serological test by standard Luminex, and standard finger stick microscopic. Their hemoglobin (Hb) and Glucose-6-Phosphate Dehydrogenase (G6PD) level will be measured. Children with Hb level<9 g/dL and/or G6PD <4 U/g Hb (male) or <6 U/g Hb (female) will be excluded. In the intervention arm (SSAT), children who are seropositive by standard Luminex and/or symptomatic LMF positive will be treated with dihydroartemisinin-piperaquine (DHA-PP) for 3 days according to national guideline and primaquine/PQ high dose (1 mg/kg BW/day for 7 days for Pv/Po, 0.25 mg/kg BW for Pf). In the control arm, children will be treated only when they show symptoms (body temperature>=36.5oC or history of fever within last 3 days) and proven positive by LMF. All treatment will be provided under direct supervision by the research team during which any adverse event/severe adverse event will be recorded. Hemoglobin level and urine will be monitored daily for 7 days of PQ administration. Post-hoc qPCR detection will be performed to determine their initial malaria status. Several additional tests will also be performed to all participants during this initial screening: microscopic examination of shallow vasculature of the ankle (light microscopy-skin/LMS), magneto-optical detection of hemozoin, and post-hoc point-of-care/POC serological test.

After enrollment, all children will be actively followed for 9 months every 4 weeks for post-hoc assessment by qPCR. Anytime during this follow up period, children becoming acutely ill will be tested for malaria by LMF, and referred to Primary Health Center to receive treatment when positive. Furthermore, household members of these infected children will also be screened for malaria infection by LMF and post-hoc LMS and qPCR. This family screening will be performed by 2x house visit (7-10 AM and 7-10 PM). Treatment will be given for those found positive by LMF regardless of their symptoms. Antimalarial treatment provided during this follow up period will be according to national standard guideline: 3 days of DHA-PP plus PQ (single 0.25 mg/kg BW dose for Pf, daily 0.25 mg/kg BW dose for 14 days for Pv/Po).

At the end of study, Pv serological test and LMF will be performed to all schoolchildren. Those found positive by LMF will be referred to Primary Health Center to receive treatment according to national standard guideline.

Sponsor: WEHI, Funding: NHMRC, Grant number: GNT1102297

ELIGIBILITY:
Inclusion Criteria:

* resident of study area and attending selected elementary school in Grade 1-5 or middle school Grade 1-3
* no evidence of health condition that would interfere with study participation
* assent of child and documented parental informed consent

Exclusion Criteria:

* G6PD deficiency as determined by SD Biosensor quantitative determination of <70% G6PD activity (<6 U/g Hb).
* Haemoglobin < 9 g/dL

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1133 (Actual)
Dates: Start 2022-02-09 (Actual); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence reduction | 9 month of follow up
  Difference of P. vivax incidence by PCR between children serologically screened and those receiving routine care.

SECONDARY OUTCOMES:
Time-to recur | 9 month
  Difference in the time-to recur of P. vivax by PCR in SSAT and control arms.
Recurrence number | 9 month
  Difference in the number of recurrent P. vivax by PCR in SSAT vs. control arms
Recurrent symptomatic P. vivax | 9 month
  Difference in the incidence of recurrent symptomatic P. vivax by microscopy in SSAT vs control arms
Seroconversion rate | 9 month
  Seroconversion rate before and after intervention in SSAT and control arms.
point-of-care assay performance | one month
  Sensitivity and specificity of point-of-care antibody detection test vs. gold standard Luminex assay
Adverse event and severe adverse event | 9 month
  Adverse event (AE) and Severe Adverse Event (SAE) of high dose PQ in schoolchildren.
Sahli Hb | One month
  Hb level in Sahli's method, Standard G6PD (SD Biosensor Inc., ROK) in comparison with (HemoCue AB, Angelholm, Sweden).
Skin gametocyte | 9 month
  Sensitivity and specificity of microscopic examination to detect parasitemia from the shallow skin vasculature of the ankle (light microscopy-skin/LMS) compared to standard microscopic (light microscopy-finger/LMF) and PCR.
Gametocyte duration | 9 month
  Mean duration time of gametocyte in LMS and LMF
Hemozoin detection | One month
  Sensitivity and specificity of magneto-optical hemozoin detection (MOD) compared to standard malaria detection and PCR.

CONTACTS AND LOCATIONS:
Overall Officials: Inge Sutanto, MD, PhD, Principal Investigator — Indonesia University
Locations (1):
- Tanjung Tiram Primary Health Center, Tanjung Tiram, Batubara, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
What data that will be shared:
  Only fully anonymized data sets will be shared as required for transparency and to fulfil publication requirements.
  Who will have access to the data:
  Researcher who provide a methodologically sound proposal.
  Where will the data be available:
  The data will be available upon request.
  When will the data be shared:
  Immediately following publication. No end date.
  How will researchers locate and access the data:
  Proposal should be sent to akosasih@eocru.org as the Study Coordinator of the trial. To gain access, data requestor will need to sign data access agreement.
Supporting Information: Study Protocol
Time Frame: No end date
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research

DOCUMENTS (1):
  • Study Protocol (2019-08-21): https://cdn.clinicaltrials.gov/large-docs/74/NCT04223674/Prot_000.pdf